CLINICAL TRIAL: NCT01516853
Title: Non-invasive Quantification of Liver Iron With MRI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0473; 2011-0473 (Other: Institutional Review Board); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison)
Record Dates: First submitted 2011-08-17; First posted 2012-01-25 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Iron Overload; Hemosiderosis
MeSH Terms: conditions — Iron Overload; Hemosiderosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patient Group: Subjects with known or suspected iron overload will undergo serum iron measurements and a non-contrast MRI scan.
  Interventions: Device: Non-contrast MRI
- Control Group: Subjects with no known history of iron overload or liver disease will undergo a serum iron measurement and a non-contrast MRI scan.
  Interventions: Device: Non-contrast MRI

INTERVENTIONS:
Device: Non-contrast MRI — Non-contrast MRI will be performed on each subject, at both 1.5T and 3.0T. Different MRI sequences (spin-echo and gradient-echo) will be used, with varying acquisition parameters (e.g., echo times, spatial resolution).

SUMMARY:
The purpose of this study is to validate magnetic resonance imaging as a biomarker of hepatic iron concentration (HIC). Excessive accumulation of iron in the body is highly toxic, specifically in the liver. Accurate, non-invasive assessment of HIC is needed for diagnosis, quantitative staging and treatment monitoring or hepatic iron overload.

DETAILED DESCRIPTION:
Excessive accumulation of iron in the body can result from abnormal intestinal absorption in hereditary hemochromatosis or repeated intravenous blood transfusions (ie: transfusional hemosiderosis). Excess body iron is highly toxic, and requires treatment aimed at reducing body iron stores. Measurement of body iron stores is critical for detection of iron overload, staging its severity and monitoring of iron-reducing therapies that are often extremely expensive (>$40,000/year) and carry their own toxicities. MRI has been shown to be very sensitive to the presence of iron. The investigators have developed an MRI-based method for rapid iron quantification (for instance, whole liver in a single breath-hold). The purpose of this work is to validate this new method using the FDA-approved Ferriscan technique (Resonance Health, Claremont, Australia) as a reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Controls: 18 years or older with no known history of iron overload or liver disease.
* Patients: 10 years or older with known or suspected iron overload

Exclusion Criteria:

* Patients with contraindications to MRI (eg. pacemaker, contraindicated metallic implants, claustrophobia, etc) and pregnant females (as determined by self-report during MRI safety screening) will be excluded.
* For control subjects, those with known liver disease will be excluded.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with known or suspected iron overload are identified and recruited in 3 different ways, 1) referral from the Division of Hematology/Oncology and Pediatric Hematology/Oncology, 2) via clinical reading of abdominal MRIs for evidence of iron overload, and 3) participants identified to have serum ferritin levels >500 by UW Hospital Clinical Laboratory will be invited to participant. Controls were recruited from a recruitment database.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Calibration Curve of Liver R2* vs. HIC Measured by FerriScan | Up to 1 day
  Accuracy of non-contrast R2*-MRI for measuring hepatic iron concentration.
Correlation of Ferritin and Liver R2* | up to 1 day
  Linear correlation between serum ferritin values and MRI R2* values
Correlation of Ferritin and HIC Measured by FerriScan | up to 1 day
  Linear correlation between serum ferritin values and FerriScan hepatic iron measurement.

SECONDARY OUTCOMES:
Variability of cardiac R2* with different imaging parameters | up to 1 day
  Robustness of Proposed Method for Cardiac R2* Estimation. Measure variability of cardiac R2* with different imaging parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Reeder, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconsin Institutes for Medical Research, Madison, Wisconsin, United States

REFERENCES:
- [Result] Hernando D, Cook RJ, Diamond C, Reeder SB. Magnetic susceptibility as a B0 field strength independent MRI biomarker of liver iron overload. Magn Reson Med. 2013 Sep;70(3):648-56. doi: 10.1002/mrm.24848. Epub 2013 Jun 25. PMID 23801540
- [Result] Sharma SD, Hernando D, Horng DE, Reeder SB. Quantitative susceptibility mapping in the abdomen as an imaging biomarker of hepatic iron overload. Magn Reson Med. 2015 Sep;74(3):673-83. doi: 10.1002/mrm.25448. Epub 2014 Sep 8. PMID 25199788
- [Result] Horng DE, Hernando D, Reeder SB. Quantification of liver fat in the presence of iron overload. J Magn Reson Imaging. 2017 Feb;45(2):428-439. doi: 10.1002/jmri.25382. Epub 2016 Jul 13. PMID 27405703